CLINICAL TRIAL: NCT05492409
Title: Extension Study of Long-term Safety and Immunogenicity of GNR-069 Patients With Idiopathic Thrombocytopenic Purpura Who Completed Phase 3 RMP-ITP-III Clinical Trial
Brief Title: Study of the Safety and Immunogenicity of Long-term GNR-069 Therapy in ITP Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AO GENERIUM (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RMP-ITP-III-X
Record Dates: First submitted 2022-08-03; First posted 2022-08-08 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-03

CONDITIONS: Idiopathic Thrombocytopenic Purpura
Keywords: Idiopathic thrombocytopenic purpura; ITP; Thrombocytopenia; Thrombocytopoiesis; Bleeding; Hemorrhagic syndrome; Petechial rash; Ecchymosis; Fc-peptide; Recombinant DNA technology; Thrombopoietin receptors; Platelet formation; Fc fragment of human immunoglobulin IgG 1; Low platelet count; ITP treatment; Platelets; Haemorrhage; Platelet destruction; Impaired thrombopoiesis; Megakaryocytes; Autoantibodies; Splenectomy; Cytotoxic; T cells; Thrombopoietin receptor agonists; Thrombopoietin receptor mimetic; TPO-RAs; romiplostim; Nplate
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Thrombocytopenia; Hemorrhage; Purpura; Ecchymosis | interventions — romiplostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GNR-069 (Experimental): Weekly subcutaneous injections of GNR-069 in the individually titrated dose.
  Interventions: Biological: GNR-069

INTERVENTIONS:
Biological: GNR-069 — Once a week as a subcutaneous injection.
  Other Names: romiplostim

SUMMARY:
It is a phase III extension study to assess safety and immunogenicity of long-term therapy with GNR-069 in patients with idiopathic thrombocytopenic purpura

DETAILED DESCRIPTION:
It is an extension study in patients with ITP who completed participation in RMP-ITP-III clinical trial.

The study will be conducted in three stages:

* Transition visit - 1 day (transition of clinical trial participants from the RMP-ITP-III study to the RMP-ITP-III-X study);
* Treatment period - minimum 26 weeks;
* Follow-up period - 1 week. Patients will then be provided with the study therapy till the product market access with only safety data collection.

ELIGIBILITY:
Inclusion Criteria:

* Completion of participation in the study RMP-ITP-III while maintaining the clinical effectiveness of romiplostim therapy

Exclusion Criteria:

* Hypersensitivity to the components of the study drug or E. Coli proteins;
* Pregnancy or breastfeeding;
* Any diseases and conditions that, in the opinion of the Investigator, may hinder the patient's participation in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2024-04-03 (Actual); Study Completion 2024-04-03 (Actual)

PRIMARY OUTCOMES:
Frequency and severity of adverse events associated with the use of the GNR-069 | up to 29 weeks
  Adverse events will be assessed based on complaints, physical examination and laboratory data.
Number of undesirable events of particular interest in the study (Bleeding;Thrombotic/thromboembolic events) | up to 29 weeks
  The event of particular interest in this study are bleeding and thrombotic/thromboembolic events of any location.
Number of clinically significant bleeding on Visits 1-5 | up to 29 weeks
  The clinically significant bleeding will be considered events ≥ grade 2 according to CTCAE 5.0.
Number and proportion of the patient with antidrug antibodies. | up to 29 weeks
  The antidrug antibodies willl be characterized by their type, titer and neutralizing activity.

SECONDARY OUTCOMES:
Frequency of the loss of the treatment response | up to 27 weeks
  Loss of the treatment response is assessed as absense of platelet increase ≥ 50,0 х 109/L on the 4 weeks treatment with maximal study drug dose.
Platelet count dynamics at Visits 1-5 | up to 5 weeks
  The platalets must be counted till week 5
Сhange in ITP-BAT bleeding scores from baseline to week 27 | up to 27 weeks
  ITP-specific bleeding assessment tool (ITP-BAT) will be calculated at baseline and at week 27.

CONTACTS AND LOCATIONS:
Overall Officials: Oksana A. Markova, MD, MSc, Study Chair — AO GENERIUM
Locations (13):
- Russia (13):
  - Federal State Budgetary Educational Institution of Higher Education "Bashkir State Medical University" of the Ministry of Health of the Russian Federation, Ufa, Bashkortostan Republic
  - State Budgetary Institution of Healthcare Irkutsk awarded the "Sign of Honor" Order Regional Clinical Hospital, Irkutsk, Irkutsk Oblast
  - State Budgetary Health Institution of the Kaluga Region "Kaluga Regional Clinical Hospital", Kaluga, Kaluga Oblast
  - State budgetary institution of health care of the Nizhny Novgorod region "Nizhny Novgorod Regional Clinical Hospital named after N. A. Semashko", Nizhny Novgorod, Nizhny Novgorod Oblast
  - Llc "Medis", Nizhny Novgorod, Nizhny Novgorod Oblast
  - Federal State Budgetary Educational Institution of Higher Education "Novosibirsk State Medical University" of the Ministry of Health of the Russian Federation, Novosibirsk, Novosibirsk Oblast
  - Federal State Budgetary Educational Institution of Higher Education "Rostov State Medical University" of the Ministry of Health of the Russian Federation, Rostov-on-Don, Rostov Oblast
  - State Health Institution of the Tula Region "Tula Regional Clinical Hospital", Tula, Tula Oblast
  - State Budgetary Institution of Healthcare of the city of Moscow "Moscow Clinical Scientific and Practical Center named after A.S. Loginov" Department of Health of the city of Moscow, Moscow
  - Federal State Budget Funded Institution National Medical Research Center of Hematology, Ministry of Health of the Russian Federation (MoH of Russia), Moscow
  - State budgetary health care institution of the city of Moscow "City Clinical Hospital named after V.V. Veresaev of the Department of Health of the City of Moscow", Moscow
  - Federal State Budgetary Institution "National Medical Research Center named after V.A. Almazov" of the Ministry of Health of the Russian Federation, Saint Petersburg
  - Municipal budgetary institution "Central City Hospital No. 7", Yekaterinburg

IPD SHARING:
Plan to Share IPD: No